CLINICAL TRIAL: NCT06601452
Title: Exploring the Biological Basis of Tonifying the Kidney and Regulating the Menstrual Cycle in the Treatment of Anovulatory Infertility Based on the Circadian Rhythm of the Biological Clock
Brief Title: Clinical Trial of Anovulatory Infertility
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Affiliated Hospital of Nanjing University of Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024NL-111-02
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovary Syndrome; Diminished Ovarian Reserve; Ovulation Disorder
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: (i) Types of trial design: Multicentre, prospective, cross-sectional study; multicentre, prospective, double-blind, randomised controlled trial.
  (II) Principles of trial design
  1. Number of cases: A total of 650 cases were included in the study, including 300 healthy women of reproductive age (divided into three groups according to age: 21-27 years old, 28-34 years old, 35-41 years old, 100 cases in each group), 150 cases of women with normal ovarian function who underwent in vitro fertilization-embryo transplantation (IVF-ET) due to male factor (divided into three groups according to age: 21-27 years old, 28-34 years old, 35-41 years old, 100 cases in each group). 34 years old, 35-41 years old, 50 cases in each group), 100 cases of PCOS infertility, 100 cases of DOR infertility.
  2. Random control: According to the accepted principles of validity, safety and comparability, SPSS 27 statistical software, define the random seed number '20240001', according to 1:1 to generate the random se
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chinese medicine treatment group（PCOS） (Experimental): Beginning on day 5 of the menstrual cycle, the treatment group was treated with a combination of Zi Yin and Yang Formula sequential treatment based on the control group, and Zi Yin and Yang Formula sequential treatment (Tuning Zhou Zi Yin Granules + Tuning Zhou and Yang Granules) was used in the 3 menstrual cycles prior to the IVF advancement week. Starting on the 5th day of the menstrual cycle, take the Tuning Zhou Zi Yin Granules (in-hospital preparation) orally. 2 packets each time, 3 times a day, 14 days of treatment; regulating Zhou Zhi Yin Granules (hospital preparation development), oral. Take 2 sachets each time, 3 times a day for 14 days.
  Interventions: Drug: a compound prescription of Chinese medicine
- Chinese medicine treatment group（DOR） (Experimental): Beginning on day 5 of the menstrual cycle, the treatment group was treated with a combination of Zi Yin and Yang Formula sequential treatment based on the control group, and Zi Yin and Yang Formula sequential treatment (Tuning Zhou Zi Yin Granules + Tuning Zhou and Yang Granules) was used in the 3 menstrual cycles prior to the IVF advancement week. Starting on the 5th day of the menstrual cycle, take the Tuning Zhou Zi Yin Granules (in-hospital preparation) orally. 2 packets each time, 3 times a day, 14 days of treatment; regulating Zhou Zhi Yin Granules (hospital preparation development), oral. Take 2 sachets each time, 3 times a day for 14 days.
  Interventions: Drug: a compound prescription of Chinese medicine

INTERVENTIONS:
Drug: a compound prescription of Chinese medicine — The enrolled patients were treated with 3 cycles of sequential treatment with Nourishing Yin and Replenishing Yang formula before entering the cycle (Tuning Weekly Nourishing Yin Granules + Tuning Weekly Replenishing Yang Granules), and the egg retrieval cycle used an antagonist regimen to obtain the eggs.

SUMMARY:
This project aims to study the expression of clock genes and related proteins in follicular fluid and granulosa cells, depicting the periodic, amplitude, and phase changes of biological clock genes and related proteins in women of different ages during the reproductive period and in patients with ovulatory disorders. The study compares the periodicity, amplitude, and phase changes of Clock/Bmal1-TTFLs-klotho related proteins and genes in PCOS, DOR patients, and age-matched women with normal ovarian function, aiming to identify the key segments of ovarian clock gene period rhythm disorder under different disease states, and screen the key time points of clock gene oscillation abnormality. Omics analysis of the differences between groups, analysis of the relationship between gene transcription translation, protein expression, metabolites, and the expression of clock genes, and deduction of the dynamic changes and interaction relationships of the biological processes within the ovaries in regulating ovulatory disorders using the method of reinforcing the kidney and regulating the menstrual cycle. This aims to clarify that maintaining the ovarian biological clock period rhythm is an important biological basis for "the kidney dominating reproduction". The regulation mechanism of the treatment of ovulatory disorders using the method of reinforcing the kidney and regulating the menstrual cycle is explained from the perspective of the ovarian biological clock period rhythm.

ELIGIBILITY:
Inclusion Criteria:

1) meet the diagnostic criteria of infertility; 2) aged between 28 and 34 years old; 3) meet the diagnostic criteria of PCOS or DOR and the Chinese medicine diagnosis is kidney deficiency, or the ovarian function is normal in the case of IVF fertilization due to the male factor; 4) assisted in fertilization with IVF-ET antagonist or microstimulation; 5) the patients can tolerate the relevant treatment of the present study, and the compliance is good; 6) they have not used any medication before the treatment and have signed the informed consent. 7) Patients who have not used any medication before the treatment and have signed the informed consent for enrollment.

Exclusion Criteria:

1) Age > 35 years old; 2) Body mass index (BMI) ≥ 25kg/m2; 3) Abnormal karyotype of either spouse; 4) Uterine infertility, such as endometrial polyps, uterine adhesions, submucosal fibroids, adenomyosis, congenital uterine anomalies, etc.; 5) Endometriosis; 6) Repeated abortion; 7) Untreated hydrosalpinx; 8) Those who had used endocrine-affecting drugs in the last three months; 9) Combination of other contraindications to assisted reproduction techniques for conception such as psychiatric disorders, severely impaired liver or kidney function, thrombotic disorders, and malignant tumors.10) Those who were unable to give full informed consent due to intellectual or behavioral disabilities.11) Suspected or confirmed history of alcohol or drug abuse.12) According to the investigator's judgment (12) Other medical conditions that, in the judgment of the investigator, reduce the likelihood of enrollment or complicate enrollment, such as frequent changes in the work environment that may result in loss of visits.13) Allergy, such as a history of allergy to two or more medications or foods, or a known allergy to the components of the medication.14) Patients participating in a clinical trial of another medication.

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 650 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Human data | Main symptoms and signs: first day of the initial consultation, the third day of the menstrual cycle without entering the treatment cycle, the day of egg collection, and 14 days after the FET are each observed and recorded once.
  Serum indicators: Serum was collected on the 3rd and 21st day of the menstrual cycle before entering the treatment cycle, and ELISA was performed to detect changes in the amount of Bmal1, Clock, klotho, Per1, Per2, Per3, Cry1, Cry2, AMH, INHB, and sex hormones (E2, FSH, LH, P, and T) in the serum.
  (2) Follicular fluid index: follicular fluid was retained on the day of ovulation, and changes in the concentration of Bmal1, Clock, klotho, AMH, INHB, and sex hormones (E2, FSH, LH, P, and T) in the follicular fluid were detected by ELISA.
  (3) Granulosa cell indexes: Ovarian granulosa cells were cultured in vitro for 24 hours on the day of egg collection, and changes in mRNA and protein of the ovarian clock genes Bmal1, Clock, klotho, Per1, Per2, Per3, Cry1 and Cry2 were detected by qPCR and WB at 3-hour intervals.
  (4) Histological indicators: follicular fluid and ovarian granulosa cells were retained on the day of egg collection for UPLC-Q-TOF/MS metabolomics, whole genome microarray genom

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China